CLINICAL TRIAL: NCT06195592
Title: The Effect of Nutritional Status of Patients Undergoing Open-Heart Surgery on The Development Postoperative Delirium
Brief Title: Development of Delirium in Patients Undergoing Open-Heart Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kubra Gunes (Other)
Responsible Party: Sponsor-Investigator, Kubra Gunes, RN, MSc, Uludag University
Organization: Uludag University (Other)
Other Study IDs: 2023-16/16
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Open-Heart Surgery
Keywords: delirium; malnutrition; open-heart surgery
MeSH Terms: conditions — Delirium; Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malnutrition is a prevalent issue among patients undergoing cardiac surgery. This can lead to delirium risk factors, including postoperative functional and cognitive impairment. Assessing the patient's nutritional status before open-heart surgery may decrease the incidence of delirium and the psychological and physiological problems associated with it. The objective of this study was to examine the relationship between nutritional status and the incidence of postoperative delirium in patients who have undergone open-heart surgery.

DETAILED DESCRIPTION:
Upon examining the literature, it was found that the incidence of delirium after open heart surgery ranged from 3% to 70% (Tomakin et al., 2020). Postoperative delirium has numerous risk factors, including predisposing and accelerating factors. Predisposing risk factors comprise malnutrition and electrolyte imbalance, cognitive impairment, depression, and other psychiatric disorders such as dementia (Velayati et al., 2019; Wilson et al., 2020). This study aims to investigate the relationship between the nutritional status of patients undergoing open heart surgery and the development of postoperative delirium. The study will be conducted in the Cardiovascular Surgery Intensive Care Unit of Bursa Uludag University Health Application and Research Centre Hospital between September 2023 and February 2024. Data will be collected using the Personal Information Form, Nutritional Risk Screening Score 2002 (NRS-2002), Delirium Risk Assessment Form, Visual Analogue Scale for Pain Levels, Richmond Agitation Sedation Scale, Glasgow Coma Scale, and Confusion Assessment Scale in Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Having undergone open heart surgery
* No mental deficiency and visual and hearing impairment
* No psychiatric diagnosis and no medication for this purpose
* Participants' acceptance to participate in the research
* The patient is not in coma (RASS score between -3 and +4, GCS score of 10 and above)

Exclusion Criteria:

* Open heart surgery under emergency conditions
* Diagnosed with delirium, dementia, psychiatric illness before surgery
* Alcohol and drug addiction
* Dying in the intensive care unit within 24 hours

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: To be eligible for the study, the patient must be at least 18 years old and have undergone open-heart surgery. They should not have any mental or sensory impairments, psychiatric diagnoses, or be taking medication for this purpose. Additionally, they should not be in a coma, with a RASS score between -3 and +4 and a GCS score of 10 or higher.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Recognising Delirium | 6 months
  Recognising delirium in malnourished patients prior to open heart surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nursel Vatansever, Principal Investigator — Uludag University
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] European Delirium Association; American Delirium Society. The DSM-5 criteria, level of arousal and delirium diagnosis: inclusiveness is safer. BMC Med. 2014 Oct 8;12:141. doi: 10.1186/s12916-014-0141-2. PMID 25300023
- [Result] Wilson JE, Mart MF, Cunningham C, Shehabi Y, Girard TD, MacLullich AMJ, Slooter AJC, Ely EW. Delirium. Nat Rev Dis Primers. 2020 Nov 12;6(1):90. doi: 10.1038/s41572-020-00223-4. PMID 33184265
- [Result] Velayati A, Vahdat Shariatpanahi M, Shahbazi E, Vahdat Shariatpanahi Z. Association between preoperative nutritional status and postoperative delirium in individuals with coronary artery bypass graft surgery: A prospective cohort study. Nutrition. 2019 Oct;66:227-232. doi: 10.1016/j.nut.2019.06.006. Epub 2019 Jun 14. PMID 31357095